CLINICAL TRIAL: NCT03849001
Title: Impact of Acute Leg Cycling at Different Intensities on Restless Legs Syndrome Severity in Persons With Multiple Sclerosis
Brief Title: Impact of Acute Leg Cycling at Various Intensities on RLS Severity in Persons With MS
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study halted prematurely, prior to enrollment of first participant
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Robert W Motl, Primary Investigator, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-300002951
Record Dates: First submitted 2019-02-19; First posted 2019-02-21 (Actual); Last update posted 2019-12-02 (Actual); Status verified 2019-11

CONDITIONS: Multiple Sclerosis; Restless Legs Syndrome
Keywords: Exercise
MeSH Terms: conditions — Multiple Sclerosis; Restless Legs Syndrome; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise Conditions (Experimental): Participants will undergo four "Exercise Conditions" (i.e., light intensity leg cycling, moderate intensity leg cycling, vigorous intensity leg cycling, and a seated, quiet rest) in a randomized, counterbalanced order.
  Interventions: Behavioral: Exercise Conditions

INTERVENTIONS:
Behavioral: Exercise Conditions — Light Exercise
Behavioral: Exercise Conditions — Moderate Exercise
Behavioral: Exercise Conditions — Vigorous Exercise
Behavioral: Exercise Conditions — Seated Rest

SUMMARY:
The purpose of this study is to evaluate the impact of acute leg cycling conditions at three different intensities versus a control condition condition on symptoms of restless legs syndrome (RLS) in persons with multiple sclerosis (MS). This study includes a proposed sample of 24 participants diagnosed with both MS and RLS that will complete four sessions of supervised exercise or rest conditions in the lab, one session per week, over the course of four weeks.

DETAILED DESCRIPTION:
The aim of this study is to evaluate the impact of acute leg cycling conditions at three different intensities (i.e., light, moderate, and vigorous) versus a control condition (i.e., quiet rest) on symptoms of RLS in persons with MS. This study involves a within-subjects, repeated measures design that includes a proposed sample of 24 participants diagnosed with both MS and RLS. Participants will complete four sessions with supervised exercise or rest conditions in the lab, one session per week, over the course of four weeks. The order of the three conditions will be randomized and counterbalanced and include: (1) leg cycling with no resistance (i.e., light), (2) leg cycling at moderate intensity, (3) leg cycling at vigorous intensity, and (4) seated, quiet rest (i.e., control condition). The primary study outcome includes the objective measure of RLS severity using the Suggested Immobilization Test (SIT) that will be administered immediately before and immediately after each condition (i.e., light, moderate, vigorous, and quiet rest).

ELIGIBILITY:
Inclusion Criteria:

* 18-54 years of age
* Diagnosis of multiple sclerosis
* Has not experienced a relapse in the last 30 days
* Positive screening for restless legs syndrome
* Restless legs syndrome severity of moderate or greater
* Ambulatory with or without an aide

Exclusion Criteria:

* Moderate or high risk for undertaking strenuous or maximal exercise
* Diagnosis of: radiculopathy, peripheral edema, peripheral neuropathy, iron deficiency (i.e., anemia), renal disease, or diabetes

Ages: 18 Years to 54 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
Restless Legs Syndrome Severity as measured by the Suggested Immobilization Test (SIT) | 10 minutes pre-exercise condition
  Participants will be reclined at a 45 degree angle on a padded treatment table with legs outstretched and will be instructed to avoid any voluntary movement of the legs for the 60 minute duration of the test. Periodic limb movements during wakefulness (PLMW) will be quantified using two accelerometers and self-reported severity of leg discomfort during the SIT will be assessed using a visual analog scale (VAS) that ranges from 0 (no discomfort) to 100 (extreme discomfort) every five minutes during the test. The SIT will be completed immediately before the light exercise condition to capture pre-exercise RLS severity.
Restless Legs Syndrome Severity as measured by the Suggested Immobilization Test (SIT) | 10 minutes post-exercise condition
  Participants will be reclined at a 45 degree angle on a padded treatment table with legs outstretched and will be instructed to avoid any voluntary movement of the legs for the 60 minute duration of the test. Periodic limb movements during wakefulness (PLMW) will be quantified using two accelerometers and self-reported severity of leg discomfort during the SIT will be assessed using a visual analog scale (VAS) that ranges from 0 (no discomfort) to 100 (extreme discomfort) every five minutes during the test. The SIT will be completed immediately after the light exercise condition to capture post-exercise RLS severity.
Restless Legs Syndrome Severity as measured by the Suggested Immobilization Test (SIT) | 10 minutes pre-exercise condition
  Participants will be reclined at a 45 degree angle on a padded treatment table with legs outstretched and will be instructed to avoid any voluntary movement of the legs for the 60 minute duration of the test. Periodic limb movements during wakefulness (PLMW) will be quantified using two accelerometers and self-reported severity of leg discomfort during the SIT will be assessed using a visual analog scale (VAS) that ranges from 0 (no discomfort) to 100 (extreme discomfort) every five minutes during the test. The SIT will be completed immediately before the moderate exercise condition to capture pre-exercise RLS severity.
Restless Legs Syndrome Severity as measured by the Suggested Immobilization Test (SIT) | 10 minutes post-exercise condition
  Participants will be reclined at a 45 degree angle on a padded treatment table with legs outstretched and will be instructed to avoid any voluntary movement of the legs for the 60 minute duration of the test. Periodic limb movements during wakefulness (PLMW) will be quantified using two accelerometers and self-reported severity of leg discomfort during the SIT will be assessed using a visual analog scale (VAS) that ranges from 0 (no discomfort) to 100 (extreme discomfort) every five minutes during the test. The SIT will be completed immediately after the moderate exercise condition to capture post-exercise RLS severity.
Restless Legs Syndrome Severity as measured by the Suggested Immobilization Test (SIT) | 10 minutes pre-exercise condition
  Participants will be reclined at a 45 degree angle on a padded treatment table with legs outstretched and will be instructed to avoid any voluntary movement of the legs for the 60 minute duration of the test. Periodic limb movements during wakefulness (PLMW) will be quantified using two accelerometers and self-reported severity of leg discomfort during the SIT will be assessed using a visual analog scale (VAS) that ranges from 0 (no discomfort) to 100 (extreme discomfort) every five minutes during the test. The SIT will be completed immediately before the vigorous exercise condition to capture pre-exercise RLS severity.
Restless Legs Syndrome Severity as measured by the Suggested Immobilization Test (SIT) | 10 minutes post-exercise condition
  Participants will be reclined at a 45 degree angle on a padded treatment table with legs outstretched and will be instructed to avoid any voluntary movement of the legs for the 60 minute duration of the test. Periodic limb movements during wakefulness (PLMW) will be quantified using two accelerometers and self-reported severity of leg discomfort during the SIT will be assessed using a visual analog scale (VAS) that ranges from 0 (no discomfort) to 100 (extreme discomfort) every five minutes during the test. The SIT will be completed immediately after the vigorous exercise condition to capture post-exercise RLS severity.
Restless Legs Syndrome Severity as measured by the Suggested Immobilization Test (SIT) | 10 minutes pre-rest (Control) condition
  Participants will be reclined at a 45 degree angle on a padded treatment table with legs outstretched and will be instructed to avoid any voluntary movement of the legs for the 60 minute duration of the test. Periodic limb movements during wakefulness (PLMW) will be quantified using two accelerometers and self-reported severity of leg discomfort during the SIT will be assessed using a visual analog scale (VAS) that ranges from 0 (no discomfort) to 100 (extreme discomfort) every five minutes during the test. The SIT will be completed immediately before the seated, quiet rest condition to capture pre-rest RLS severity.
Restless Legs Syndrome Severity as measured by the Suggested Immobilization Test (SIT) | 10 minutes post-rest (Control) condition
  Participants will be reclined at a 45 degree angle on a padded treatment table with legs outstretched and will be instructed to avoid any voluntary movement of the legs for the 60 minute duration of the test. Periodic limb movements during wakefulness (PLMW) will be quantified using two accelerometers and self-reported severity of leg discomfort during the SIT will be assessed using a visual analog scale (VAS) that ranges from 0 (no discomfort) to 100 (extreme discomfort) every five minutes during the test. The SIT will be completed immediately after the seated, quiet rest condition to capture post-rest RLS severity.

SECONDARY OUTCOMES:
Restless Legs Syndrome Severity as measured by the International Restless Legs Syndrome Study Group Scale (IRLS) | Baseline through screening
  In order to characterize RLS symptom severity over the previous week, participants will be asked to complete the IRLS. The IRLS is a validated 10-question survey that provides a global score commonly used to assess the overall severity of symptoms as well as the frequency and impact of symptoms on daily life in reference to the previous week. Overall symptom severity scores are determined by combining the sum of the answers on the questionnaire with with a range of 0 to 40 and higher scores indicating greater severity of symptoms.
Restless Legs Syndrome Severity as measured by the International Restless Legs Syndrome Study Group Scale (IRLS) | Baseline through week 1
  In order to characterize RLS symptom severity over the previous week, participants will be asked to complete the IRLS. The IRLS is a validated 10-question survey that provides a global score commonly used to assess the overall severity of symptoms as well as the frequency and impact of symptoms on daily life in reference to the previous week. Overall symptom severity scores are determined by combining the sum of the answers on the questionnaire with with a range of 0 to 40 and higher scores indicating greater severity of symptoms.
Restless Legs Syndrome Severity as measured by the International Restless Legs Syndrome Study Group Scale (IRLS) | week 1 through week 2
  In order to characterize RLS symptom severity over the previous week, participants will be asked to complete the IRLS. The IRLS is a validated 10-question survey that provides a global score commonly used to assess the overall severity of symptoms as well as the frequency and impact of symptoms on daily life in reference to the previous week. Overall symptom severity scores are determined by combining the sum of the answers on the questionnaire with with a range of 0 to 40 and higher scores indicating greater severity of symptoms.
Restless Legs Syndrome Severity as measured by the International Restless Legs Syndrome Study Group Scale (IRLS) | week 2 through week 3
  In order to characterize RLS symptom severity over the previous week, participants will be asked to complete the IRLS. The IRLS is a validated 10-question survey that provides a global score commonly used to assess the overall severity of symptoms as well as the frequency and impact of symptoms on daily life in reference to the previous week. Overall symptom severity scores are determined by combining the sum of the answers on the questionnaire with with a range of 0 to 40 and higher scores indicating greater severity of symptoms.
Restless Legs Syndrome Severity as measured by the International Restless Legs Syndrome Study Group Scale (IRLS) | week 3 through week 4
  In order to characterize RLS symptom severity over the previous week, participants will be asked to complete the IRLS. The IRLS is a validated 10-question survey that provides a global score commonly used to assess the overall severity of symptoms as well as the frequency and impact of symptoms on daily life in reference to the previous week. Overall symptom severity scores are determined by combining the sum of the answers on the questionnaire with with a range of 0 to 40 and higher scores indicating greater severity of symptoms.
Restless Legs Syndrome Severity as measured by the International Restless Legs Syndrome Study Group Scale (IRLS) | week 4 through week 5
  In order to characterize RLS symptom severity over the previous week, participants will be asked to complete the IRLS. The IRLS is a validated 10-question survey that provides a global score commonly used to assess the overall severity of symptoms as well as the frequency and impact of symptoms on daily life in reference to the previous week. Overall symptom severity scores are determined by combining the sum of the answers on the questionnaire with with a range of 0 to 40 and higher scores indicating greater severity of symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Robert W Motl, PhD, Principal Investigator — University of Alabama at Birmingham

IPD SHARING:
Plan to Share IPD: No